CLINICAL TRIAL: NCT00780988
Title: A Pilot Study to Assess the Safety and Feasibility of Autologous Tumor Cell-TLR9 Agonist Vaccination Prior to Autologous Hematopoietic and Immune Cell Rescue in Metastatic Colorectal Cancer
Brief Title: Feasibility of Autologous Tumor Cell-TLR9 Agonist Vaccination for Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-09112008-1298; COR0008
Record Dates: First submitted 2008-10-23; First posted 2008-10-28 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Neoplasms; Anal, Colon, and Rectal Cancers
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Transplantation

INTERVENTIONS:
Biological: Autologous tumor cell + CpG vaccine
Procedure: Autologous hematopoietic and immune cell rescue (transplantation)

SUMMARY:
Current therapies for metastatic colorectal cancer only prolong life for approximately 2 years. A more innovative therapy that prolongs life significantly or even cures is needed. Bone marrow transplantation is a curative therapy for patients with leukemias and lymphomas. Tumor eradication in the case of transplantation of the patient's own marrow (autologous transplantation) is based on the intensive chemotherapy and/or radiotherapy used for conditioning. Tumor eradication in the case of transplantation using the marrow of a normal donor is based on both tumor reduction from conditioning and the immune elimination of tumor cells by T cells in the donor transplant that recognize the foreign tissue antigens expressed by the tumor cells and kill these cells. The use of bone marrow transplantation to treat tumors other than leukemia and lymphoma has been limited, and studies of transplantation of the patient's own marrow for the treatment of advanced /metastatic breast cancer have not conclusively shown benefit beyond conventional therapy.

Recently, the Strober lab developed a preclinical model that effectively treated colon cancer in mice by combining immunotherapy and autologous bone marrow transplantation in order to markedly augment the anti-tumor potency of immunotherapy. They used the CT26 colon cancer as the therapeutic target either as a single subcutaneous tumor nodule, as a disseminated tumor in the lungs and peritoneum, or as a metastatic tumor in the liver depending on the route of administration of the tumor cells in BALB/c mice. Mice were vaccinated mice with established primary tumors or disseminated/ metastatic disease with irradiated tumor cells mixed with the adjuvant CpG, and found that vaccination alone had no effect on tumor growth. Similarly radiation conditioning of tumor bearing hosts followed by transplantation of bone marrow and spleen cells or purified T cells and hematopoietic stem cells from unvaccinated donors of the same strain had no effect. In contrast, radiation conditioning of mice followed by transplantation of hematopoietic and immune cells from donors of the same strain vaccinated with tumor cells and CpG cured almost all subcutaneous primary as well as disseminated and metastatic tumors in the hosts. A similar result was obtained after autologous transplantation of hematopoietic and immune cells from tumor bearing mice that had been vaccinated after tumor establishment. Investigation of tumor infiltrating cells showed that the injected donor T cells do not accumulate in the tumors unless the host has been irradiated before injection.

Based on this model, we have assembled a team of Stanford University faculty members with expertise in gastrointestinal cancers, immunotherapy, radiation oncology, and bone marrow transplantation in the Departments of Medicine and Pathology to translate the preclinical findings into a Phase I safety and feasibility clinical study for the treatment of 10 patients with metastatic colorectal cancer. Resected tumor cells will be irradiated and mixed with CpG to create a vaccine. Patients will receive subcutaneous vaccination at weeks 1 and 2 after resection. Six weeks later, immune T cells and then G-CSF "mobilized" purified blood progenitor cells will be harvested from the blood and cryopreserved. If needed patients will receive chemotherapy for tumor reduction. When disease is controlled off chemotherapy, patients will receive a conditioning regimen of fludarabine (30mg/m2 daily x 3 days) followed by intensive fractionated total body irradiation. The dose of fTBI will be escalated using a 3+3 design to ensure safety and will range from 400 to 800 gray. The patient will then undergo hematopoietic and immune cell rescue. They will undergo a third vaccination within 7-14 days after transplant. Thereafter, serial monitoring of tumor burden will continue.

Immune monitoring will occur before and after vaccination as well as after transplantation. Tests will include in vitro anti-tumor immune responses of T cells (proliferation, cytotoxicity, cytokine secretion etc.) to stimulation with whole tumor cells and tumor cell lysates pulsed on to antigen presenting cells, anti-tumor antibody responses, and immune reconstitution after transplantation.

DETAILED DESCRIPTION:
As the third most common cancer in incidence and second in mortality, colorectal cancer (CRC) significantly impacts the lives of many Americans.1 In 2008, it is estimated that 148,810 cases will be diagnosed and 49,960 patients will die from this disease. Approximately 20% of patients present with metastatic disease at diagnosis. The introduction of more effective chemotherapy regimens and biologically targeted agents over the last few years has led to considerable improvement in treatment options for metastatic CRC yet median survival approximates only 2 years. Resection of the primary tumor when clinically indicated followed by combinations of oxaliplatin or irinotecan with intravenous or oral 5-FU, leucovorin, and bevacizumab for first-line therapy of metastatic CRC is standard of care.

In 2004, Goldberg and colleagues established FOLFOX4 as the standard of care chemotherapy regimen in metastatic CRC when they demonstrated its superiority over two older regimens, IFL (bolus 5-FU/leucovorin/irinotecan) and IROX (irinotecan/oxaliplatin), in terms of prolonging median overall survival (OS), progression-free survival (PFS), and increased response.2 FOLFOX4 increased median survival time to 19.5 months compared to 15 months and 17.4 months for IFL and IROX respectively (p= .0001; HR .66, 95% CI 0.54-0.82). Time to progression was also significantly increased to 8.7 months compared to 6.9 and 6.5 months (p=.0014). Furthermore FOLFOX-4 effected a 45% overall response rate compared to 31% (p=.002) and 35% (p=.03) for IFL and IROX respectively. It also induced significantly less associated grade; 3 nausea, vomiting, diarrhea, febrile neutropenia, and dehydration than the other two regimens.

Hoping to improve this regimen further, capecitabine, an oral pro-drug of 5-FU, was introduced. It has significant advantages over infusional 5-FU including ease of administration with its oral formulation, lack of infusion-related toxicities, and decreased duration of hospitalization and clinic time. Multiple trials have pitted capecitabine-based therapies against infusional 5-FU regimens and have shown comparable efficacy.3-8 Overall toxicity profiles are also comparable between the two regimens with the exception of less myelosuppression and more hand-foot syndrome with capecitabine compared to the infusional-5-FU-based regimens. Thus, in clinical practice, CAPOX (capecitabine-oxaliplatin) is largely considered to be a comparable regimen to FOLFOX, with significantly more convenient administration.

The addition of targeted therapies that inhibit vascular endothelial growth factor (VEGF) and endothelial growth factor receptor (EGFR) to the 5-FU/LV regimens have further increased survival. Bevacizumab, a monoclonal antibody against VEGF, was approved for metastatic CRC in 2004 after the pivotal phase III trial, AVF2107g, showed a significant improvement in OS from 15.6 months to 20.3 months (HR for death, 0.66, p <0.001) with the addition of bevacizumab to IFL.9 PFS and response were also significantly increased from 6.2 months to 10.6 months (p<0.001) and 34.8% to 44.8% (p= 0.004) respectively. The first phase III trial to evaluate the combination of bevacizumab with oxaliplatin-based chemotherapy (FOLFOX-4 or CAPOX), NO16966, demonstrated that the addition of bevacizumab improved PFS by 1.4 months (9.4 vs. 8.0 months, HR 0.83, p=.0023) but overall response rates were similar.10 Median OS also increased from 19.9 months in the placebo group to 21.3 months in the bevacizumab arm but was not statistically significant (HR 0.89, p=.077).

Cetuximab, a mouse/human chimeric monoclonal antibody to EGFR, has also shown promise in metastatic CRC.11, 12 The BOND trial, a multicenter randomized phase II trial showed a significant doubling of response rate and a 2.6 month increase in PFS with the combination of irinotecan-cetuximab over cetuximab alone in the second line setting, but no difference in median OS.11 These results led the FDA to approve cetuximab in February 2004 for second-line treatment either as a monotherapy in those who cannot tolerate irinotecan or in combination with irinotecan in those who do not have a response to irinotecan alone. The CRYSTAL trial, a phase III multicenter randomized trial also demonstrated that cetuximab holds promise in the first line setting.13 In this trial (n=1217), the addition of cetuximab to FOLFIRI significantly increased response rate by 6% (46.9% vs. 38.7%, p=0.005) and PFS by 1.9 months (p=0.036). Trials evaluating the first line use of cetuximab with oxaliplatin-based regimens appear promising and are ongoing.14, 15 When using cetuximab, the presence of K-RAS mutations must be considered. Activating mutations in the K-RAS gene are present in 40-45% of colorectal cancer patients.16 The presence of these mutations correlates with a worse outcome and a lack of response to cetuximab in patients with advanced chemotherapy-refractory CRC.17, 18 Even with these new agents and improved combinations, median survival for metastatic CRC patients remains less than 2 years with less than 5%surviving to 5 years.19 Furthermore, one can expect 20% of patients to progress within 4-6 months.10 Better regimens and treatments are greatly needed to impact this pervasive and fatal disease.

ELIGIBILITY:
Inclusion Criteria:- Histologically confirmed Stage IV, TxNxM1 colon adenocarcinoma with a surgically accessible primary or metastatic site.

* Estimated survival of 6 months or greater
* Primary may be in place
* Age 18-70
* Must have an ECOG performance status of 0 or 1
* Must have adequate organ and marrow function. Specifically:

  * Absolute neutrophil count (ANC) > 1500/uL
  * Platelet count >= 100 x 109/L
  * Total bilirubin <= 2.0 x the upper limit of normal (ULN)
  * Alkaline phosphatase, AST, and/or ALT <2.5 x the ULN for patients
  * without evidence of liver metastases; <5 X ULN for patients with
  * documented liver metastases
  * Serum creatinine < 2.0 mg/dL
  * Hemoglobin > 9 g/dL

    a. Patients may be transfused or receive epoetin alfa to maintain or exceed this level up to the hemoglobin level recommended on the current label for epoetin alfa. There is concern that hemoglobin levels greater than the level recommended by the current labeling have been associated with the potential increased risk of thrombotic events and increased mortality. Also, a rapid increase in hemoglobin may exacerbate hypertension (a concern in patients with pre-existing hypertension and if bevacizumab is administered).
  * Cardiac ejection fraction >40 % by transthoracic echo or MUGA scan within 12 wks of transplant
  * Adequate pulmonary function tests (PFTs) within 6 wks of transplant

    a. DLCO >=60% predicted
  * Patients must be HIV negative
* No prior therapy which would preclude the use of total body irradiation
* Pathology must be reviewed and diagnosis confirmed by Stanford University Medical Center
* Ability to understand and the willingness to sign a written informed consent document.
* Ability and capacity to comply with the study and follow-up procedures.; Exclusion Criteria:- Disease-Specific Exclusions

  * Radiotherapy within 28 days prior to the day of tumor resection (Day 1).
  * No myelosuppressive chemotherapy within 28 days prior to the day of tumor resection
  * History of brain metastases, regardless if treated.
* Co-morbid diseases or intercurrent illness

  * Active infection or fever > 38.5°C within 3 days of starting treatment
  * History of other malignancies within 5 years prior to Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma, squamous-cell carcinoma of the skin, carcinoma in situ of the cervix, early-stage bladder cancer, or low-grade endometrial cancer
  * Malignancies that have undergone a putative surgical cure (i.e., localized prostate cancer post-prostatectomy) within 5 years prior to Day 1 may be discussed with the Medical Monitor.
  * History or presence of autoimmune disorders requiring treatment
  * Any other medical conditions (including mental illness or substance abuse) deemed by the clinician to be likely to interfere with a patient's ability to provide informed consent, cooperate, or participate in the study, or to interfere with the interpretation of the results.
  * Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
  * Any prior history of hypertensive crisis or hypertensive encephalopathy
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix A)
  * History of myocardial infarction or unstable angina within 6 months prior to study enrollment
  * History of stroke or transient ischemic attack within 6 months prior to study enrollment
  * Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
  * Symptomatic peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy that is not intentionally pharmacologically-induced Serious, non-healing wound, ulcer, or bone fracture
  * Proteinuria at screening as demonstrated by either:

    1. Urine protein: creatinine (UPC) ratio >= 1.0 at screening OR
    2. Urine dipstick for proteinuria >= 2+ (patients discovered to have >=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate <= 1g of protein in 24 hours to be eligible).
* Radiation-specific exclusions

  o Prior radiation to >25% of the marrow
* Pregnancy

  * Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control.

    a. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days of study entry.
  * Nursing patients will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of using an autologous tumor cell vaccine in combination with standard chemotherapy followed by investigational autologous hematopoietic and immune cell rescue in terms of acceptable clinical toxicity.

SECONDARY OUTCOMES:
Preliminary efficacy in terms of response and time to progression
Ex vivo analysis of immune response

CONTACTS AND LOCATIONS:
Overall Officials: George Albert Fisher M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States